CLINICAL TRIAL: NCT02602379
Title: Evaluation of NoL Index and ANI Variations After Nociceptive Stimulation Under Different Rates of Infusion of Intravenous Remifentanil in Patients Undergoing Laparotomies With Intraoperative Epidural Analgesia
Brief Title: Evaluation of NoL Index and ANI After Nociceptive Stimulation at Different Infusion Rates of Remifentanil Infusion
Status: Completed | Type: Observational
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Medasense Biometrics Ltd (Other)
Responsible Party: Principal Investigator, Philippe Richebé, MD, PhD, Professor of anesthesiology, Maisonneuve-Rosemont Hospital
Other Study IDs: HMR14090
Record Dates: First submitted 2015-10-25; First posted 2015-11-11 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Pain
Keywords: Pain; Monitoring; Analgesia Nociception Index; NoL; Nociception Level; Remifentanil
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Tetanic stimulation: Single arm study. See Study description for a through description of the intervention.
  Interventions: Other: Tetanic stimulation

INTERVENTIONS:
Other: Tetanic stimulation — Standard Tetanic stimulation will be used as the stimulus to evaluate responses of the intraoperative pain indexes (ANI and NoL) at different concentration of i.v. remifentanil during anesthesia.

SUMMARY:
Contrary to "immobility" and, to a lesser extent, to the "hypnosis/unconsciousness" component of general anaesthesia, the monitoring of "analgesia" remains largely elusive, evaluated mainly through poorly sensitive and potentially undesirable changes in patients' vital signs. This has led the industry to pursue the development of various devices and indices based on other physiological parameters such as heart rate variability (HRV), electroencephalogram (EEG), skin conductance, to name only a few. To the best of the knowledge, none of these parameters on its own has shown sufficient capacity in detecting different degrees of pain/analgesia balance to gain wide clinical use.

The purpose of this prospective observational study is to evaluate the response of a single-parameter index (the Analgesia Nociception Index [ANI]) and a multi-parameter index (the Nociception Level [NoL] Index) when patients under combined general anaesthesia/epidural anaesthesia for laparotomies are subjected to a standardized painful stimulus (a tetanic stimulation over the ulnar nerve at 70 mA, 100 Hz for 30 seconds) at different doses of remifentanil infusion at steady state (0,005 mcg/kg/min; 0,05 mcg/kg/min; 0,1 mcg/kg/min; 0,15 mcg/kg/min). With the painful stimulus held constant but the analgesia provided gradually increased, it is expected to characterize the response of these two indices to different levels of nociception/anti-nociception balance.

DETAILED DESCRIPTION:
Patients scheduled for elective abdominal surgery by laparotomy (general surgery or gynaecological surgery) will receive a thoracic epidural (around T9-T10/T10-T11) and general anesthesia. Apart from standard monitoring, the ANI (derived from the EKG) and the NoL index (obtained via a finger probe) will be recorded. The epidural catheter will be injected with 6-10 ml of lidocaine 2% with epinephrine 5 mcg/ml to produce anesthetic level of neuraxial blocade and then be perfused with the same solution at 4-8 ml/hour. After incision and confirmation of adequate blocade with the epidural local anesthetic, the patient will receive a series of painful electric stimulation with a standard nerve stimulator applied over the ulnar nerve in tetanic mode for 30 seconds at 100 Hz and 70mA. Each stimulation will occur at a different rate of infusion of IV remifentanil at steady state (0,005 mcg/kg/min; 0,05 mcg/kg/min; 0,1 mcg/kg/min; 0,15 mcg/kg/min). A stimulation at 0,005 mcg/kg/min will be done before and after epidural loading with local anesthetics to look for altered variations in analysed parameters. The variation and the kinetic of the variations after stimulations will be observed for heart rate, mean blood pressure, BIS, ANI and NoL index.

ELIGIBILITY:
Inclusion Criteria:

* ASA status I, II or III
* Elective abdominal surgery with median laparotomy under general anaesthesia and epidural analgesia.

Exclusion Criteria:

* Coronary artery disease
* Serious cardiac arrhythmias (including atrial fibrillation)
* Patient refusal
* History of substance abuse
* Chronic use of psychotropic and/or opioid drugs
* Use of drugs that act on the autonomic nervous system (including β-blockers)
* History of psychiatric diseases or psychological problems
* Contraindications to epidural analgesia
* Allergy to remifentanil
* Unexpected difficult airway requesting excessive, possibly painful airway manipulations.
* Dural puncture during epidural catheter installation
* Failure of epidural analgesia
* Surgical unexpected complications requiring strong haemodynamic support (transfusions, vasopressors, inotropes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective abdominal surgery by laparotomy (general surgery or gynaecological surgery) who will receive a thoracic epidural (around T9-T10/T10-T11) and general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Correlation between NoL index responses to electrical stimulus and the i.v. doses of remifentanil infusion given during anesthesia. The n of patients (40 in this study) is calculated on this primary outcome. | At time of surgery
  The electrical stimulus will be applied on the forearm of the asleep patient at different doses of iv remifentanil (0.005mcg/kg/min to a maximum of 0.15 mcg/kg.min during anesthesia for abdominal surgery with active intraoperative epidural pain management). It will be evaluated whether or not exists a correlation between the doses of iv remifentanil and the responses of the Nol index after electrical stimulus.

SECONDARY OUTCOMES:
NoL index changes after a standardized electrical stimulus at 4 different concentrations of iv remifentanil infusion | At time of surgery
  Measure the NoL changes after a nociceptive stimulus at various intravenous remifentanil infusion doses.
ANI index changes after a standardized electrical stimulus at 4 different concentrations of iv remifentanil infusion | At time of surgery
  Measure the ANI changes after a nociceptive stimulus at various intravenous remifentanil infusion doses. ANI being another uniparametric pain index.
Heart rate changes after a standardized electrical stimulus at 4 different concentrations of iv remifentanil infusion | At time of surgery
  Measure the changes of Heart Rate after a nociceptive stimulus at various intravenous remifentanil infusion doses.
Mean Blood Pressure changes after a standardized electrical stimulus at 4 different concentrations of iv remifentanil infusion | At time of surgery
  Measure the changes of Heart Rate after a nociceptive stimulus at various intravenous remifentanil infusion doses.
Sensitivity and specificity of NoL index, ANI index, Heart Rate and Mean blood Pressure in detecting a painful stimulus such as intubation as well as standardized electrical stimulus at remifentanil infusion of 0.005 msg/kg/min | At time of surgery
  Measure the sensitivity and specificity of these 4 criteria in detecting a painful stimulus such as intubation and standardized electrical stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Richebé, M.D. PhD, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada